#### Free and Informed Consent Form - Electronic Version

Evaluation of the effectiveness of a multicomponent nature-based intervention for well-being and relationship with nature in different natural areas: a randomized clinical trial.

# Free and Informed Consent Form Participants aged > 18 years


#### Introduction

You are being invited to voluntarily participate in the study entitled "Evaluation of the effectiveness of a multicomponent nature-based intervention for well-being and relationship with nature in different natural areas: a randomized clinical trial". For you to decide to be part of it, you will need to know what your participation consists of, as well as the possibilities of risks and benefits and confirm your participation by signing this free and informed consent form.

If you have any questions, after or while reading this term, please feel free to talk to the researcher responsible for conducting the study and who can clarify your doubts.

The decision to take part in the study is voluntary and you may refuse to participate or withdraw from the study at any time without any consequences whatsoever to you.

The objective of this research is to verify how an intervention in the middle of nature influences or not your well-being, your vitality, happiness, and we want to know how is the relationship you have with nature.

If you agree to participate in this research, you will participate in two stages: (1) Welcome, presentation of the project team, explanation about the research objectives, about interventions, about the instruments to be completed and about the random possibility of be included in the Control Group (CG) or Intervention Group (IG). So, if you agree to participate, you must express your agreement by signing this Free and Informed Consent Form (ICF) in person but in electronic format; (2) Completion of the questionnaires: sociodemographic and environmental characterization, Scale of connection with nature, Engagement with nature, Scale of well-being, Scale of self-

perception of happiness, Scale of vitality, Scale of empathy with animals, Scale of compassion, with an estimated time of 20 to 30 minutes.

Then, you will be directed to one of the two groups, according to a draw performed by a *software*: Group 1, in which you will take a light walk, of approximately one hour, accompanied by a researcher throughout the trail, but you will not have interactions with him, except when filling out the questionnaires. If you are drawn into this group, you will be guided to perceive nature through the senses (Hearing, vision, smell, touch); Group 2, which will take the same light walk, in the same stretch of Group 1, also with the same duration of approximately one hour, however, the researcher will offer more targeted information about plants and animals of the place, show some birds that are in the path and will provide guidance for appreciatively looking at the surrounding nature and experiencing it through the senses. In this Group 2, we will also ask that during the 30 days following the walk you continue to observe nature, following our Inspiration Guide and Eco challenges Guide, and make records on our *Instagram* or profile - @umtempocomenatureza, using the *hashtag* #ecochallenge.


At the end of the walk, you will answer the Well-being Scale, Self-Perception of Happiness Scale and Vitality Scale again, participating in both Group 1 and Group 2, which should last from 10 to 20 minutes. Thus, to participate in this research you need to have up to two hours of availability at the time of the walk, at a single time.

Also, 30 days after this walk, we will send you a link by email that will provide us with the answer to the third and last moment of filling out the following questionnaires: Scale of connection with nature, Engagement with nature, Scale of good -being, Self-Perception of Happiness Scale, Vitality Scale, lasting 20 to 30 minutes.

## Participant's duties

In order to carry out this study, it is important that you answer all the questionnaires at the three times indicated above, however you have the right not to answer any question, without the need for explanation or justification for doing so.

## Risks and inconveniences

This research brings some risks related to the environment in which the study is developed. As it is a natural area, there is a risk of being bitten by an insect or other type of animal present in the region. Therefore, the place where you will walk has already been previously analyzed by the study team, with smooth and clean terrain to avoid these risks and will always be accompanied by specialists who will promptly identify any potential risk situation, as they are experienced in these places. Even so, should something happen, you will be entitled to full assistance free of charge due to direct/indirect and immediate/delayed damages, for as long as necessary. There is also the risk of some embarrassment to a question that is more sensitive to you personally. There is minimal risk of breach of confidentiality and confidentiality of any invasion of the institutional platform where the data will be stored.


## **Study Benefit**

If the intervention in the nature of any of the groups proves to be effective, you will already be able to observe immediate effects on your well-being and your participation can help in the implementation of this activity, coming to benefit other people or even yourself in other opportunities.

## Participant rights

Your participation is voluntary and you can withdraw your consent or discontinue your participation at any time, if you prefer, without penalty and/or prejudice of any nature.

You will have access to the questions only after you have given your consent, as well as the guarantee that you have the right to access the content of the questionnaires (topics that will be addressed) before answering the questions, so that you can make your decision. in an informed manner.

Study staff will provide you with a snack to eat after your participation. There will be no remuneration for your participation and no financial reimbursement for transport expenses, since you are already in the park for your leisure and have decided to voluntarily participate in the study.

By signing this term, you do not waive any legal rights, including the right to seek compensation in the event of damage resulting from your participation.

If it is of interest to you, you may request information about the results of this study at any time when the analyzes are complete.

## **Damage**


If an injury or any damage occurs as a result of your participation in this research, full assistance will be available at no cost to you, for as long as necessary.

## Confidentiality

The study team will have access to your data, however, your anonymity is guaranteed and possible scientific publications resulting from this study will not identify you under any circumstances as a participant. The data obtained will be treated under strict confidentiality conditions.

### **Ethic**

This study was approved by the Research Ethics Committee (CEP), a group of people that ensures the protection of research participants and evaluates studies involving human beings at our institution.

This term has two copies, one being the responsible researcher and the other, duly signed by the researcher, will be sent to the email you provide to the study team.

For any ethical questions and/or related to the rights of the research participant, contact the Research Ethics Committee of Hospital Albert Einstein by phone (11) 2151-3729, or by e-mail cep@einstein.br. The Committee works from Monday to Friday, from 7 am to 5 pm and is located at Av. Albert Einstein, 627 – 2nd ss of Bloco A- Morumbi – São Paulo – SP - 05652-900.

For any questions related to the study, please feel free to contact those responsible for conducting the study, Eliseth Leão, by telephone: +55 (11) 2151-1032 or +55 (11) 996186489, or by e-mail: <a href="mailto:enatureza@einstein.br">enatureza@einstein.br</a> or <a href="mailto:eliseth.leao@einstein.br">eliseth.leao@einstein.br</a>.

Complaints, compliments and suggestions may be sent to the Customer Service System (SAC) by calling (11) 2151-0222 or using the form identified as "contact us", available on the clinical research page, or in person.

| I have been informed of all details related to the study in which I will participate and will |
|---|
| have access to the study after accepting this electronic consent form. |
| ( ) I accept to participate in the study at Unit |
| ( ) I do not accept to participate in the study |

Pag 5/5